CLINICAL TRIAL: NCT03280823
Title: Effect of Platelet Storage on Complement Activation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shimaa Abdeleem (Other)
Responsible Party: Sponsor-Investigator, Shimaa Abdeleem, Doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: platelets and complement
Record Dates: First submitted 2017-08-29; First posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Platelet Storage
Keywords: complement system

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Platelet units are stored and complement factors are evaluated

DETAILED DESCRIPTION:
Ten units of platelets will be selected from the regular inventory of the Central Blood Transfusion Services/Assiut University Hospitals . All units of platelets will be collected, processed, and tested following the standard procedures.

Thesis units will be stored on a platelet rotator with the temperature controlled between 22 and 24c. Samples will be obtained using a sterile technique .

The investigators will take basal sample and samples on day 2,3,4 and 5. Complement components will be assayed : C4 (classical pathway), C3 (common pathway) and C5 (terminal pathway).

This evaluation will be done using ELISA technique

ELIGIBILITY:
Inclusion Criteria:

* Negative screening and confirmatory tests will be done for all platelet donors

Exclusion Criteria:

* Use of aspirin or non steroidal anti-inflammatory drugs or medication affecting the platelets.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Gender Based: Yes — Negative screening and confirmatory tests will be done for all platelet donors
Study Population: No Use of aspirin or non steroidal anti-inflammatory drugs or medication affecting the platelets.
  Negative screening and confirmatory tests will be done for all platelet donors
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Platelets can be used after storage upto 5 days instead of using in the same day of donation without complement activation. | 5 days

REFERENCES:
- [Background] Chen J, Losos M, Yang S, Li J, Wu H, Cataland S. Increased complement activation during platelet storage. Transfusion. 2017 Sep;57(9):2182-2188. doi: 10.1111/trf.14215. Epub 2017 Jul 3. PMID 28671303